CLINICAL TRIAL: NCT02361060
Title: Effects of Neuromuscular Block Reversal With Sugammadex vs Neostigmine on Postoperative Respiratory Outcomes After Major Abdominal Surgery - A Randomized Controlled Trial
Brief Title: Effects of Neuromuscular Block Reversal With Sugammadex vs Neostigmine on Postoperative Respiratory Outcomes After Major Abdominal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Enrique Alday Muñoz (Other)
Responsible Party: Sponsor-Investigator, Enrique Alday Muñoz, Principal investigator., Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Organization: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRIN-SUGAR-2014
Record Dates: First submitted 2014-12-23; First posted 2015-02-11 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Major Abdominal Surgery
MeSH Terms: interventions — Neostigmine; Sugammadex; Atropine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugammadex (Experimental): sugammadex 4 mg/kg
  Interventions: Drug: Sugammadex
- Neostigmine + Atropine (Active Comparator): Neostigmine 40µg/kg in combination with atropine 10µg/kg.
  Interventions: Drug: Neostigmine; Drug: Atropine

INTERVENTIONS:
Drug: Neostigmine — 40mcg/kg
  Arms: Neostigmine + Atropine
Drug: Sugammadex — 4mg/kg
  Arms: Sugammadex
Drug: Atropine — 10 mcg/kg
  Arms: Neostigmine + Atropine

SUMMARY:
Pulmonary complications are relatively frequent after surgery, and can be associated with an increase in morbidity and mortality. Although there are several causative mechanisms that can lead to postoperative pulmonary complications, alterations in the shape and motion of the chest wall are of primary importance.

In the investigator´s institution the incidence of postoperatory hypoxemia defined as pO2/FiO2 <300 is over 20% for patients after major abdominal surgery.

Observational and randomized clinical trials have demonstrated that incomplete neuromuscular recovery during the early postoperative period may result in acute respiratory events (hypoxemia and airway obstruction) and an increased risk of postoperative pulmonary complications.

A recent study in laparoscopic bariatric surgery showed that patients in which neuromuscular block reversal was done with sugammadex had less chest X-ray pathological changes than those from an historical cohort reversed with neostigmine.

The hypothesis is that differences in pulmonary complications, as atelectasis and hypoxemia, between patients reverted with sugammadex or neostigmine may be more apparent with more sensitive techniques like spirometry or lung ultrasound when they exist.

Lung ultrasound (LUS) has demonstrated a sensitivity of 90% and a specificity of 98%, to detect alveolar consolidation in critical ill patients while chest radiography data are known to be imprecise.The investigator would like to explore the utility of LUS in postsurgical patients and the relationship between degree of hypoxemia and consolidation area.

Objectives:

1. Primary: Forced vital capacity decreases after surgery. This reduction may be relieved in the absence of residual neuromuscular block. Objective is to assess differences after reversal with neostigmine versus sugammadex in:

   • Forced vital capacity (FVC)
2. Secondary objectives: To assess differences after reversal with neostigmine versus sugammadex in:

   * Atelectasis size determined by lung ultrasound (Plannimetry)
   * pO2/FiO2 <300 1 hour after surgery
   * Explore the accuracy of lung ultrasound (LUS) to diagnosis postoperative atelectasis and its correlation with chest Xray, FVC and pO2/FiO2.

Hypotheses:

1. Sugammadex NMB reversal results in a lower reduction of forced vital capacity (FVC) as compared to NMB reversal with neostigmine.
2. Atelectasis is common after major surgery. Size of atelectasis determined by lung ultrasound planimetry is lower one hour after sugammadex reversal as compared to the neostigmine group.
3. The incidence of post-surgical hypoxemia is lower in the sugammadex group as compared to the neostigmine group (Hypoxemia defined as pO2/FiO2 less than 300 is expected in 20% of patients after major abdominal surgery).
4. Lung ultrasound has a better capacity to detect alveolar consolidation than Chest Xray after major surgery.
5. Atelectasis size determine by planimetry has a good correlation with pO2/FiO2 and decrease of FVC after surgery

ELIGIBILITY:
Inclusion Criteria:

* Every patient scheduled for major abdominal surgery (liver resection, pancreatectomy, gastrectomy or any type of colectomy) will be nominated to participate in the study.
* Informed consent will be asked for after their admission to the hospital the day before the surgery.
* Patients with postoperative epidural analgesia.

Exclusion Criteria:

* Refusal to participate.
* Entry to postoperative recovery unit under mechanical ventilation.
* Hypersensitivity reactions to any of the drugs.
* Severe asthma and mild asthma under treatment.
* Myocardial infarction or coronary occlusion three months prior to surgery.
* Myasthenia gravis.
* Emergency surgery.
* Pulmonary fibrosis or very severe chronic obstructive lung disease (GOLD IV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2015-02; Primary Completion 2016-07-04 (Actual); Study Completion 2016-07-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in FVC at 1h after surgery | Basal and one hour after surgery

SECONDARY OUTCOMES:
Atelectasis size determined by lung ultrasound (Plannimetry) | One hour after surgery
Atelectasis size determined by lung ultrasound (Plannimetry) | 24 hours after surgery
pO2/FiO2 <300 | 1 hour after surgery
Asociation between atelectasis size and FVC | 1 hour after surgery
  Atelectasis size (sqr cm) will me measured by planimetry
Asociation between atelectasis size and FVC | 24 hour after surgery
  Atelectasis size (sqr cm) will me measured by planimetry
Asociation between atelectasis size and pO2/FiO2 | 1 hour after surgery
  Atelectasis size (sqr cm) will me measured by planimetry
Asociation between atelectasis size and pO2/FiO2 | 24 hour after surgery
  Atelectasis size (sqr cm) will me measured by planimetry

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Anesthesiology Service. Hospital Universitario La Princesa, Madrid, Madrid
  - Hospital Universitario de La Princesa, Madrid, Madrid

REFERENCES:
- [Background] Flockton EA, Mastronardi P, Hunter JM, Gomar C, Mirakhur RK, Aguilera L, Giunta FG, Meistelman C, Prins ME. Reversal of rocuronium-induced neuromuscular block with sugammadex is faster than reversal of cisatracurium-induced block with neostigmine. Br J Anaesth. 2008 May;100(5):622-30. doi: 10.1093/bja/aen037. Epub 2008 Apr 2. PMID 18385265
- [Background] Jones RK, Caldwell JE, Brull SJ, Soto RG. Reversal of profound rocuronium-induced blockade with sugammadex: a randomized comparison with neostigmine. Anesthesiology. 2008 Nov;109(5):816-24. doi: 10.1097/ALN.0b013e31818a3fee. PMID 18946293
- [Background] Lee C, Jahr JS, Candiotti KA, Warriner B, Zornow MH, Naguib M. Reversal of profound neuromuscular block by sugammadex administered three minutes after rocuronium: a comparison with spontaneous recovery from succinylcholine. Anesthesiology. 2009 May;110(5):1020-5. doi: 10.1097/ALN.0b013e31819dabb0. PMID 19387176
- [Background] Staals LM, Snoeck MM, Driessen JJ, Flockton EA, Heeringa M, Hunter JM. Multicentre, parallel-group, comparative trial evaluating the efficacy and safety of sugammadex in patients with end-stage renal failure or normal renal function. Br J Anaesth. 2008 Oct;101(4):492-7. doi: 10.1093/bja/aen216. Epub 2008 Jul 23. PMID 18653492
- [Background] Dahl V, Pendeville PE, Hollmann MW, Heier T, Abels EA, Blobner M. Safety and efficacy of sugammadex for the reversal of rocuronium-induced neuromuscular blockade in cardiac patients undergoing noncardiac surgery. Eur J Anaesthesiol. 2009 Oct;26(10):874-84. doi: 10.1097/EJA.0b013e32832c605b. PMID 19455040
- [Background] Yang LP, Keam SJ. Sugammadex: a review of its use in anaesthetic practice. Drugs. 2009;69(7):919-42. doi: 10.2165/00003495-200969070-00008. PMID 19441874
- [Background] Abrishami A, Ho J, Wong J, Yin L, Chung F. Sugammadex, a selective reversal medication for preventing postoperative residual neuromuscular blockade. Cochrane Database Syst Rev. 2009 Oct 7;(4):CD007362. doi: 10.1002/14651858.CD007362.pub2. PMID 19821409
- [Background] Ferreyra G, Long Y, Ranieri VM. Respiratory complications after major surgery. Curr Opin Crit Care. 2009 Aug;15(4):342-8. doi: 10.1097/MCC.0b013e32832e0669. PMID 19542885
- [Background] Squadrone V, Coha M, Cerutti E, Schellino MM, Biolino P, Occella P, Belloni G, Vilianis G, Fiore G, Cavallo F, Ranieri VM; Piedmont Intensive Care Units Network (PICUN). Continuous positive airway pressure for treatment of postoperative hypoxemia: a randomized controlled trial. JAMA. 2005 Feb 2;293(5):589-95. doi: 10.1001/jama.293.5.589. PMID 15687314
- [Background] Yu CJ, Yang PC, Wu HD, Chang DB, Kuo SH, Luh KT. Ultrasound study in unilateral hemithorax opacification. Image comparison with computed tomography. Am Rev Respir Dis. 1993 Feb;147(2):430-4. doi: 10.1164/ajrccm/147.2.430. PMID 8430970
- [Background] Murphy GS, Brull SJ. Residual neuromuscular block: lessons unlearned. Part I: definitions, incidence, and adverse physiologic effects of residual neuromuscular block. Anesth Analg. 2010 Jul;111(1):120-8. doi: 10.1213/ANE.0b013e3181da832d. Epub 2010 May 4. PMID 20442260
- [Background] Tusman G, Bohm SH, Warner DO, Sprung J. Atelectasis and perioperative pulmonary complications in high-risk patients. Curr Opin Anaesthesiol. 2012 Feb;25(1):1-10. doi: 10.1097/ACO.0b013e32834dd1eb. PMID 22113182
- See also: Sugammadex and anaphylaxis in the operating theater. — http://dx.doi.org/10.1016/j.redar.2014.02.005
- See also: Postoperative respiratory outcomes in laparoscopic bariatric surgery: Comparison of a prospective group of patients whose neuromuscular blockade was reverted with sugammadex and a his-torical one reverted with neostigmine — http://dx.doi.org/10.1016/j.redar.2013.11.009